CLINICAL TRIAL: NCT02247167
Title: Endothelial Dysfunction and Oxidative Stress in Children With Sleep Disordered Breathing.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Violi, Full professor of Internal Medicine, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: Sapienza-sdb; C26A13W4AK (Other: Sapienza University)
Record Dates: First submitted 2014-07-09; First posted 2014-09-23 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Obstructive Sleep Apnea of Child
Keywords: obstructive sleep apnoea, oxidative stress, FMD
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- adenotonsillectomy (AT) (Experimental): Children with SDB studied before and after before adenotonsillectomy.
  Interventions: Procedure: adenotonsillectomy

INTERVENTIONS:
Procedure: adenotonsillectomy — adenotonsillectomy in children with OSAS and adenotonsillar hypertrophy.

SUMMARY:
Sleep disordered breathing (SDB) is a common disease in both adults and children and is caused by the obstruction of the upper airway during sleep. Unlike adults, most cases of paediatric SDB are due to the presence of enlarged tonsils and adenoids, thus the main treatment option is adenotonsillectomy (AT). It is well known that obstructive sleep apnoea (OSA) in adults increases the risk for hypertension, coronary artery disease and stroke, and there is now mounting evidence that SDB also has a significant impact on the cardiovascular system in children with reports of elevated blood pressure, endothelial dysfunction and altered autonomic cardiovascular control.

Oxidative stress seems to play a pivotal role in impairing flow-mediated dilation (FMD) and consequently enhancing cardiovascular risk in SDB patients but the underlying mechanism is still undefined.

Previously, we demonstrated that endothelial dysfunction is directly related to NADPH oxidase activation. Furthermore, recently we assessed the association between OSA, endothelial dysfunction and oxidative stress in adults showing that increased NADPH oxidase-generated oxidative stress and arterial dysfunction are partially reversed by nasal continuous positive airway pressure treatment.

There is evidence in literature that cardiovascular morbidities associated with SDB are potentially reversible in children; AT may have a significant role in reversing the cardiovascular sequelae of SDB (e.g. children with OSA).

Nowadays, there aren't studies that analyzed the role of NADPH oxidase-generated oxidative stress in SDB children.

The purpose of the current research project is to examine the role of NADPH oxidase activity, oxidative stress, inflammation and endothelial function in SDB children, understanding the mechanisms involved in this disease.

Furthermore we will analyse the effect of a AT on inflammation, oxidative stress, NADPH oxidase activity and endothelial function in SDB children.

DETAILED DESCRIPTION:
Sleep disordered breathing (SDB) is a spectrum of diseases ranging from primary snoring to obstructive sleep apnoea (OSA). Recent studies suggested that the prevalence of SDB childhood was 7.4%. In patients with OSA, there are intermittent episodes of complete or partial obstruction leading to intermittent desaturations and/or arousals. This would result in either stimulation of sympathetic system or suppression of the vagal tone that may persist beyond sleep. The disturbance of the autonomic nervous system would result in significant changes in the cardiovascular system. The process of intermittent hypoxaemia and subsequent re-oxygenation also damages the endothelium because of the generation of free radicals. Furthermore, the excessive negative intra-thoracic pressure swing generated during the obstruction would also affect cardiac functions. In adults, OSA has been well documented to be associated with cardiovascular abnormalities such as hypertension, ischaemic heart disease, arrhythmia and heart failure.

Oxidative stress plays a crucial role in the initiation and progression of atherosclerosis. In particular, an imbalance between superoxide and nitric oxide production could be responsible for endothelial dysfunction, a key point for atherosclerotic process. Several oxidative stress-generating enzymes, including myeloperoxidase, xanthine oxidase and nicotinamide adenine dinucleotide phosphate (NADPH) may be implicated in arterial dysfunction; NADPH oxidase represents, in human, the most important source of cellular superoxide anion production. Experimental studies performed in animal models suggest a pivotal role of NADPH oxidase in modulating arterial tone. In particular, overexpression of gp91phox (NOX2), potentiates the hemodynamic response to angiotensin II. Furthermore, individuals with impaired dilation show an overexpression of the NADPH oxidase subunit p47phox in endothelial cells.

Previously, we demonstrated that endothelial dysfunction is directly related to NADPH oxidase activation; in particular we demonstrated that in patients with NADPH oxidase subunits deletion, as chronic granulomatous disease, the oxidative stress is lower and flow-mediate dilation is higher, compared to controls. Conversely, in other diseases characterized by high rate of cardiovascular events (OSAS, Peripheral arterial disease, metabolic syndrome, obesity and hypercholesterolemia), we found an endothelial dysfunction and a NOX2 overexpression.

Recently, we assessed the association between OSAS, endothelial dysfunction and oxidative stress in adults. Interestingly, the results of our study indicated that patients with OSAS have increased NOX2-generated oxidative stress and arterial dysfunction that are partially reversed by nasal continuous positive airway pressure (nCPAP) treatment.

There is evidence in literature that cardiovascular morbidities associated with SDB are potentially reversible in children; AT may have a significant role in reversing the cardiovascular sequelae of SDB (e.g. children affected by OSA).

The purpose of the current research project is to examine NADPH oxidase activity, oxidative stress, inflammation and endothelial function in children with SDB.

Expected outcomes and their interest in advances in the frontier of knowledge and their potential impact:

1. understand the mechanisms mediated by inflammation and oxidative stress involved in SDB
2. the assessment of NADPH oxidase activity could be a useful tool to identify SDB patients at high risk of cardiovascular events in order to prevent their dramatic complications.
3. Analyse the effect of a surgical correction (e.g. adenotonsillectomy) on inflammation, oxidative stress, NADPH oxidase activity and endothelial function in children; adenotonsillectomy could represent a potential therapeutic option to reduce the high cardiovascular risk of SDB children.

The study will be divided in 2 phases: a cross-sectional and an interventional study.

1. In the cross-sectional study we will include at least 100 children (50 SDB children with SDB and 50 controls), assessing markers of oxidative stress (serum isoprostanes), NADPH oxidase activity, inflammation, endothelial function (by flow-mediated dilation, FMD) and the carotid intima media thickness (IMT) measurement.
2. In the interventional study we will include at least 10 with OSA and adenotonsillar hypertrophy that will undergo to adenotonsillectomy, evaluating markers of oxidative stress (serum isoprostanes), NADPH oxidase activity, inflammation and endothelial function before and after (at least 30 days) the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

Children with diagnosed sleep breathing disorders

Exclusion Criteria:

* epilepsy
* acute or chronic cardiorespiratory or neuromuscular diseases
* chronic inflammatory diseases
* liver insufficiency
* serious renal disorders
* smoking
* vitamin assumption

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Assessment of flow mediated dilation (fmd) | Baseline, week 4

SECONDARY OUTCOMES:
Assessment of isoprostanes 8 Iso-pgf2alpha (pg/ml) levels | Baseline, 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Violi, MD, Principal Investigator — Sapienza University; Marzia Duse, MD, Study Director — Sapienza University
Locations (1):
- Sapienza University of Rome, I Clinica Medica, Research Tower, Rome, Italy

REFERENCES:
- [Background] Del Ben M, Fabiani M, Loffredo L, Polimeni L, Carnevale R, Baratta F, Brunori M, Albanese F, Augelletti T, Violi F, Angelico F. Oxidative stress mediated arterial dysfunction in patients with obstructive sleep apnoea and the effect of continuous positive airway pressure treatment. BMC Pulm Med. 2012 Jul 23;12:36. doi: 10.1186/1471-2466-12-36. PMID 22824065
- [Background] Loffredo L, Martino F, Carnevale R, Pignatelli P, Catasca E, Perri L, Calabrese CM, Palumbo MM, Baratta F, Del Ben M, Angelico F, Violi F. Obesity and hypercholesterolemia are associated with NOX2 generated oxidative stress and arterial dysfunction. J Pediatr. 2012 Dec;161(6):1004-9. doi: 10.1016/j.jpeds.2012.05.042. Epub 2012 Jun 23. PMID 22727869
- [Background] Violi F, Sanguigni V, Carnevale R, Plebani A, Rossi P, Finocchi A, Pignata C, De Mattia D, Martire B, Pietrogrande MC, Martino S, Gambineri E, Soresina AR, Pignatelli P, Martino F, Basili S, Loffredo L. Hereditary deficiency of gp91(phox) is associated with enhanced arterial dilatation: results of a multicenter study. Circulation. 2009 Oct 20;120(16):1616-22. doi: 10.1161/CIRCULATIONAHA.109.877191. Epub 2009 Oct 5. PMID 19805647
- [Derived] Loffredo L, Zicari AM, Occasi F, Perri L, Carnevale R, Angelico F, Del Ben M, Martino F, Nocella C, Savastano V, Cesoni Marcelli A, Duse M, Violi F. Endothelial dysfunction and oxidative stress in children with sleep disordered breathing: role of NADPH oxidase. Atherosclerosis. 2015 May;240(1):222-7. doi: 10.1016/j.atherosclerosis.2015.03.024. Epub 2015 Mar 18. PMID 25805361